CLINICAL TRIAL: NCT02983513
Title: Early Intervention in Preterm Infants: Effects of a Parental Training Program on Neonatal Brain Development, Visual Functions and Neurobehavioral Outcome
Brief Title: Early Intervention in Preterm Infants: Short and Long Term Developmental Outcome After a Parental Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MITP Preterm
Record Dates: First submitted 2016-11-16; First posted 2016-12-06 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Premature Birth
Keywords: Early intervention; Brain Development; Neurodevelopment
MeSH Terms: conditions — Premature Birth | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention (Experimental): The early intervention program is delivered during the NICU stay, according to the MITP and Premie Start Protocol, in order to train parents to: recognize signs of infant stress and alert-available behavior to promote mother-infant interaction; adopt principles of graded stimulation; optimize interactions and avoid overwhelming infants through facilitation strategies (for example, engage and support the visual attention of the newborn). The program is held in eight main sessions and one additional post-discharge session.
  In addition parents are trained and invited to daily promote preterm baby massage therapy and visual attention according to a detailed protocol.
  Interventions: Behavioral: Early Intervention
- Standard Care (No Intervention): Standard Care according to NICU protocols including Kangaroo Mother Care, nesting and minimal handling

INTERVENTIONS:
Behavioral: Early Intervention
  Arms: Early Intervention

SUMMARY:
Preterm infants, during their stay in the Neonatal Intensive Care Unit (NICU), face a period of stressful environment, which may negatively impact early brain development and subsequent neurobehavioral outcomes. This study aims to assess the effectiveness of training parents in reducing stressful experiences early in life and in enhancing brain development and long term developmental outcomes.

DETAILED DESCRIPTION:
Very preterm birth is associated with motor, cognitive and behavioral problems.

Micro-structural brain abnormalities, even in the absence of focal lesions, have been documented by neuroimaging studies in preterm infants at term corrected age and later in childhood. These alterations in brain maturation occurring during the neonatal period may be implicated in long-term neurobehavioral disorders later experienced by preterm babies.

However, there is increasing evidence that also negative environmental factors (intensive care, excessive sensory stimulation, paucity of parental contact etc.) can affect later outcomes.

Potential benefits of early dyadic interaction and preterm baby massage in reducing the effects of the NICU stressor environment have been demonstrated. More recently, few studies have investigated visual function in preterm infants focusing on the potential role of early visual interaction to enhance attention and improve later neurodevelopment.

The role of early intervention strategies to improve neurodevelopment has been recently emphasized.

Early intervention programs based on the concept of "individualized care" have proved to be effective in promoting brain maturation and neurodevelopmental outcome. In this context, early interventions as the Mother Infant Transaction Program (MITP) and the Premie Start, both targeting parenting, have the greatest potential to have sustained effects on child development.

In addition, recent studies have shown that exposure to stressful events in the neonatal period can cause epigenetic modifications in children born preterm; in particular alteration of serotonergic tone was observed, associated with methylation of the serotonin transporter gene, which could be implicated in the etiology of behavioral disorders observed in these children. In animal models these epigenetic effects appear to be influenced by maternal care that can epigenetically modulate the offsprings' stress response.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 25+0 and 29+6 weeks

Exclusion Criteria:

* major brain lesions as documented by cranial ultrasound (intraventricular hemorrhage > 2 grade, cystic periventricular leukomalacia)
* neurosensorial deficits (retinopathy of prematurity > stage 2)
* genetic syndromes and/or major congenital malformations
* major neonatal comorbidities

Mothers are selected according to the following inclusion criteria: age over 18 years, good comprehension of Italian language, no obvious cognitive impairments or psychiatric disorders, no drug addiction and no single-parent families.

Ages: 25 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2014-04; Primary Completion 2017-04 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Visual Assessment Battery to evaluate visual function | 40 weeks postmenstrual age
  Neonatal Visual Function is assessed using the Visual Assessment Battery developed by Ricci et al. The assessment evaluates the following items: Ocular spontaneous motility, ability to fix and follow a target, reaction to colour, visual acuity and visual attention at distance. Each item is scored as normal (score 0) or abnormal (score 1). The global score is then calculated as the sum of all the individual items, as designed by the authors.
Neonatal Behavior | 2 months corrected age
  Neonatal behavior is assessed using the Neonatal Behavior Assessment Scale that evaluates: habituation, social-interactive, motor system, state organization and regulation, autonomic system, reflexes.

SECONDARY OUTCOMES:
Brain development | 40 weeks postmenstrual age
  Conventional and advanced MRI
Developmental outcome | 24 months corrected age
  Children development is assessed using the Bayley Scales of Infant and Toddlers (Third edition) - including: cognitive, motor, language, social-emotional and adaptive behavior)
Epigenetic changes | up to 48 weeks gestational age
  epigenetic analysis is performed at birth on a cord blood sample (0.5 ml) and at hospital discharge on a peripheral blood sample (0.5 ml) collected according routine clinical procedures
overall duration of hospitalisation | up to 48 weeks gestational age
  number of days from admission to home discharge from NICU
Weight (in grams) at 40 weeks postmenstrual age | 40 week gestational age
Length(in centimeters) at 40 weeks postmenstrual age | 40 week gestational age
Head circumference (in centimeters) at 40 weeks postmenstrual age | 40 week gestational age
Acquisition of full oral feeding | up to 48 weeks gestational age
  Postmenstrual age at the acquisition of full oral feeding
Feeding with Human milk | up to 40 weeks gestational age
  Feeding with human milk at 40 weeks postmenstrual age (yes or no)
Neurodevelopmental outcome | 5-6 years of age
  Children neurodevelopment is assessed using the Griffiths Development Scales (GMDS).
  Scores range from 50 to 150 General quotient mean 100 SD 12, sub scales mean 100 SD 16 Higher scores mean a better outcome
Behavioral outcome | 5-6 years of age
  Children behavior is assessed using the Child Behavior Checklist. A T score above 70 is considered to be in the clinical range, a T score between 65 an 70 is considered borderline while a T score below 65 is considered normal
Neuromotor outcome | 5-6 years of age
  Children neuromotor is assessed using the Movement Assessment Battery for Children (Movement ABC).
  A score above 67 is considered to be in the normal range, a score between 57 an 67 is considered borderline while a score below 56 is considered pathological
Attention outcome | 5-6 years of age
  Child attention abilities is assessed using the Early Childhood Attention Battery (ECAB).
  Scaled scores range from 1 to 19. Lower scores indicate worst outcome
L1 promoter methylation levels on buccal swab | 5-6 years of age
  epigenetic analysis - L1 promoter methylation (Percent) assessment is performed on a buccal swab collected at follow-up assessment at 5-6 years.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Fumagalli, MD, Principal Investigator — Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico
Locations (1):
- NICU, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
individual patient consent would be required according to the EU GDPR and Italian regulations

REFERENCES:
- [Background] Newnham CA, Milgrom J, Skouteris H. Effectiveness of a modified Mother-Infant Transaction Program on outcomes for preterm infants from 3 to 24 months of age. Infant Behav Dev. 2009 Jan;32(1):17-26. doi: 10.1016/j.infbeh.2008.09.004. Epub 2008 Nov 20. PMID 19026450
- [Background] Provenzi L, Fumagalli M, Sirgiovanni I, Giorda R, Pozzoli U, Morandi F, Beri S, Menozzi G, Mosca F, Borgatti R, Montirosso R. Pain-related stress during the Neonatal Intensive Care Unit stay and SLC6A4 methylation in very preterm infants. Front Behav Neurosci. 2015 Apr 21;9:99. doi: 10.3389/fnbeh.2015.00099. eCollection 2015. PMID 25941480
- [Background] Guzzetta A, D'Acunto MG, Carotenuto M, Berardi N, Bancale A, Biagioni E, Boldrini A, Ghirri P, Maffei L, Cioni G. The effects of preterm infant massage on brain electrical activity. Dev Med Child Neurol. 2011 Sep;53 Suppl 4:46-51. doi: 10.1111/j.1469-8749.2011.04065.x. PMID 21950394
- [Background] Ricci D, Cesarini L, Romeo DM, Gallini F, Serrao F, Groppo M, De Carli A, Cota F, Lepore D, Molle F, Ratiglia R, De Carolis MP, Mosca F, Romagnoli C, Guzzetta F, Cowan F, Ramenghi LA, Mercuri E. Visual function at 35 and 40 weeks' postmenstrual age in low-risk preterm infants. Pediatrics. 2008 Dec;122(6):e1193-8. doi: 10.1542/peds.2008-1888. PMID 19047222
- [Background] Ricci D, Romeo DM, Serrao F, Cesarini L, Gallini F, Cota F, Leone D, Zuppa AA, Romagnoli C, Cowan F, Mercuri E. Application of a neonatal assessment of visual function in a population of low risk full-term newborn. Early Hum Dev. 2008 Apr;84(4):277-80. doi: 10.1016/j.earlhumdev.2007.10.002. Epub 2007 Nov 8. PMID 17996405
- [Derived] Fontana C, Provitera L, Bonfanti C, Schiavolin P, Polimeni B, Marasca F, Pesenti N, Iuliano R, Gangi S, Bodega B, Fumagalli M. Neurodevelopmental outcome at 5 to 6 years of age of an early intervention program in preterm infants. Sci Rep. 2025 Dec 2;15(1):45786. doi: 10.1038/s41598-025-28564-8. PMID 41331309
- [Derived] Fontana C, Marasca F, Provitera L, Mancinelli S, Pesenti N, Sinha S, Passera S, Abrignani S, Mosca F, Lodato S, Bodega B, Fumagalli M. Early maternal care restores LINE-1 methylation and enhances neurodevelopment in preterm infants. BMC Med. 2021 Feb 5;19(1):42. doi: 10.1186/s12916-020-01896-0. PMID 33541338
- [Derived] Fontana C, De Carli A, Ricci D, Dessimone F, Passera S, Pesenti N, Bonzini M, Bassi L, Squarcina L, Cinnante C, Mosca F, Fumagalli M. Effects of Early Intervention on Visual Function in Preterm Infants: A Randomized Controlled Trial. Front Pediatr. 2020 Jun 4;8:291. doi: 10.3389/fped.2020.00291. eCollection 2020. PMID 32582595